CLINICAL TRIAL: NCT03036150
Title: A Study to Evaluate the Effect of Dapagliflozin on Renal Outcomes and Cardiovascular Mortality in Patients With Chronic Kidney Disease
Acronym: Dapa-CKD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D169AC00001; 2016-003896-24 (EudraCT Number)
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease (CKD); Cardiovascular Events (CV); Phase III outcome trial
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Patients will be randomized 1:1 to either dapagliflozin or placebo.
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo matching dapagliflozin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg or 5 mg tablets given once daily, per oral use.
  Other Names: Forxiga TM; Farxiga TM
  Arms: Dapagliflozin
Drug: Placebo — Placebo matching dapagliflozin 10 mg or 5 mg
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of dapagliflozin on renal outcomes and cardiovascular mortality in patients with chronic kidney disease.

DETAILED DESCRIPTION:
This is an international, multicentre, event-driven, randomized, double-blind, parallel group, placebo-controlled study, evaluating the effect of dapagliflozin versus placebo, given once daily in addition to standard of care, to prevent the progression of chronic kidney disease (CKD) or cardiovascular (CV)/renal death.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent prior to any study specific procedures
* Female or male aged ≥18 years at the time of consent
* eGFR ≥25 and ≤75 mL/min/1.73m2 (CKD-EPI Formula) at visit 1
* Evidence of increased albuminuria 3 months or more before visit 1 and UACR ≥200 and ≤5000 mg/g at visit 1
* Stable, and for the patient maximum tolerated labelled daily dose, treatment with ACE-I or ARB for at least 4 weeks before visit 1, if not medically contraindicated,

Exclusion Criteria:

* Autosomal dominant or autosomal recessive polycystic kidney disease, lupus nephritis or ANCA-associated vasculitis
* Receiving cytotoxic therapy, immunosuppressive therapy or other immunotherapy for primary or secondary renal disease within 6 months prior to enrolment
* History of organ transplantation
* Receiving therapy with an SGLT2 inhibitor within 8 weeks prior to enrolment or previous intolerance of an SGLT2 inhibitor
* Type 1 diabetes mellitus
* New York Heart Association (NYHA) class IV Congestive Heart Failure at the time of enrolment
* MI, unstable angina, stroke or transient ischemic attack within 12 weeks prior to enrolment

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4304 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (309):
- United States (49):
  - Research Site, Birmingham, Alabama
  - Research Site, Hawaiian Gardens, California
  - Research Site, Lomita, California
  - Research Site, Los Angeles, California
  - Research Site, Palo Alto, California
  - Research Site, San Dimas, California
  - Research Site, San Ramon, California
  - Research Site, Vista, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Boynton Beach, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Naples, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Topeka, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Metairie, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, Albany, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Jersey Shore, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greer, South Carolina
  - Research Site, Kingsport, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Odessa, Texas
  - Research Site, Burke, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Tacoma, Washington
- Argentina (14):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad Autonoma Buenos Aires
  - Research Site, Ciudad Autonoma de Buenos Aire
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Mar del Plata
  - Research Site, Nueve de Julio
  - Research Site, Rosario
  - Research Site, San Luis
  - Research Site, San Miguel de Tucumán
  - Research Site, San Nicolás
  - Research Site, Santa Fe
  - Research Site, Santa Rosa
- Brazil (10):
  - Research Site, Botucatu
  - Research Site, Campinas
  - Research Site, Caxias do Sul
  - Research Site, Curitiba
  - Research Site, Joinville
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (19):
  - Research Site, Edmonton, Alberta
  - Research Site, Red Deer, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Concord, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Smiths Falls, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Gatineau, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Sherbrooke, Quebec
- China (23):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Foshan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Jilin
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanjin
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shengyang
  - Research Site, Shenzhen
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Yinchuan
  - Research Site, Yueyang
- Denmark (6):
  - Research Site, Aarhus
  - Research Site, Gentofte Municipality
  - Research Site, Herlev
  - Research Site, Hillerød
  - Research Site, København Ø
  - Research Site, Roskilde
- Germany (14):
  - Research Site, Aschaffenburg
  - Research Site, Bad Oeynhausen
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Hanover
  - Research Site, Magdeburg
  - Research Site, München
  - Research Site, Münster
  - Research Site, Schweinfurt
  - Research Site, Tübingen
  - Research Site, Ulm
- Hungary (9):
  - Research Site, Budapest
  - Research Site, Eger
  - Research Site, Gyula
  - Research Site, Kistarcsa
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Velence
- India (16):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Calicut
  - Research Site, Chennai
  - Research Site, Ernākulam
  - Research Site, Hyderabad
  - Research Site, Kanpur
  - Research Site, Kolkata
  - Research Site, Lucknow
  - Research Site, Madurai
  - Research Site, Maharashtra
  - Research Site, Mangalore
  - Research Site, Nagpur
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Vijayawada
- Japan (41):
  - Research Site, Amagasaki-shi
  - Research Site, Asahikawa-shi
  - Research Site, Beppu-shi
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Daito-shi
  - Research Site, Fujisawa-shi
  - Research Site, Fukuoka
  - Research Site, Higashiibaraki-gun
  - Research Site, Iizuka-shi
  - Research Site, Itabashi-ku
  - Research Site, Kamakura-shi
  - Research Site, Kanazawa
  - Research Site, Kawachinagano-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kobe
  - Research Site, Koga-shi
  - Research Site, Koshigaya-shi
  - Research Site, Kumamoto
  - Research Site, Kurashiki
  - Research Site, Matsumoto-shi
  - Research Site, Nagano
  - Research Site, Nagoya
  - Research Site, Naha
  - Research Site, Neyagawa
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Sapporo
  - Research Site, Shizuoka
  - Research Site, Takarazuka-shi
  - Research Site, Toride-shi
  - Research Site, Tsu
  - Research Site, Tsuchiura-shi
  - Research Site, Ueda-shi
  - Research Site, Uji-shi
  - Research Site, Yaizu-shi
  - Research Site, Yokohama
- Mexico (11):
  - Research Site, Aguascalientes
  - Research Site, Cuernavaca
  - Research Site, Culiacán
  - Research Site, D.F
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, Mazatlán
  - Research Site, México
  - Research Site, Minatitlán
  - Research Site, Monterrey
  - Research Site, Saltillo
- Peru (9):
  - Research Site, Arequipa
  - Research Site, Callao
  - Research Site, Chorrillos
  - Research Site, Cusco
  - Research Site, Ica
  - Research Site, Lima
  - Research Site, Piura
  - Research Site, San Isidro
  - Research Site, San Miguel
- Philippines (9):
  - Research Site, Bacolod
  - Research Site, Cebu
  - Research Site, Cebu City
  - Research Site, Dasmariñas
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Makati City
  - Research Site, Marikina City
  - Research Site, Quezon City
- Poland (16):
  - Research Site, Bielsko-Biala
  - Research Site, Bochnia
  - Research Site, Chorzów
  - Research Site, Ciechanów
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Legnica
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Oława
  - Research Site, Poznan
  - Research Site, Ruda Śląska
  - Research Site, Rzeszów
  - Research Site, Szczecin
  - Research Site, Tczew
- Russia (16):
  - Research Site, Chelyabinsk
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Perm
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Tver'
  - Research Site, Ufa
  - Research Site, Vladikavkaz
  - Research Site, Volgograd
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- South Korea (9):
  - Research Site, Ansan-si
  - Research Site, Deagu
  - Research Site, Goyang-si
  - Research Site, Gwangju
  - Research Site, Jeonju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Uijeongbu-si
  - Research Site, Wŏnju
- Spain (9):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Burela (Lugo)
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Malmo
  - Research Site, Stockholm
  - Research Site, Uppsala
- Ukraine (13):
  - Research Site, Cherkasy
  - Research Site, Chernivtsі
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv Region
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Rivne
  - Research Site, Ternopil
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
- United Kingdom (8):
  - Research Site, Cardiff
  - Research Site, Glasgow
  - Research Site, Hull
  - Research Site, Kent
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Salford
  - Research Site, Swansea
- Vietnam (4):
  - Research Site, Biên Hòa
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heerspink HJL, Chertow GM, Rossing P, Correa-Rotter R, Sjostrom CD, Toto RD, Wheeler DC, Jongs N. Effects of Dapagliflozin on Progression of CKD According to Different Rates of Pretrial eGFR Loss. Clin J Am Soc Nephrol. 2025 Nov 1;20(11):1527-1535. doi: 10.2215/CJN.0000000810. Epub 2025 Sep 9. PMID 41128261
- [Derived] Bakker WM, Heerspink HJL, Jongs N, Correa-Rotter R, Rossing P, Toto RD, Wheeler DC, McMurray JJV, Langkilde AM, Gansevoort RT, Chertow GM, Vart P. Effects of Dapagliflozin on Health-Related Quality of Life in Patients with CKD. J Am Soc Nephrol. 2026 Jan 1;37(1):101-109. doi: 10.1681/ASN.0000000776. Epub 2025 Jul 18. PMID 40679863
- [Derived] Oshima M, Buizen L, Jongs N, Levin A, Chertow GM, Wheeler DC, Heerspink HJL, Arnott C, Jardine MJ, Mahaffey KW, Pollock C, Herrington WG, Perkovic V, Neuen BL. Sodium-Glucose Cotransporter 2 Inhibition and Hospitalizations in Patients with CKD: A Meta-Analysis of Kidney Outcome Trials. Clin J Am Soc Nephrol. 2025 Jul 14;20(9):1206-1214. doi: 10.2215/CJN.0000000771. PMID 40658498
- [Derived] Jongs N, Gasparyan SB, Frison L, Schloemer P, Brinker M, Little DJ, Heerspink HJL. Use of eGFR Slope Thresholds as End Point Components in a Kidney Disease Progression Hierarchical Composite End Point. J Am Soc Nephrol. 2025 Dec 1;36(12):2421-2430. doi: 10.1681/ASN.0000000766. Epub 2025 Jun 17. PMID 40526444
- [Derived] van Mil D, Vart P, Chertow GM, Gansevoort RT, Rossing P, Toto RD, Correa-Rotter R, Langkilde AM, Sjostrom CD, Wheeler DC, Heerspink HJL. Baseline, Early Changes, and Residual Albuminuria: Post Hoc Analysis of a Randomized Clinical Trial of Dapagliflozin in Chronic Kidney Disease. Clin J Am Soc Nephrol. 2024 Dec 1;19(12):1574-1584. doi: 10.2215/CJN.0000000000000550. PMID 39475817
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Zhang Z, Heerspink HJL, Chertow GM, Correa-Rotter R, Gasparrini A, Jongs N, Langkilde AM, McMurray JJV, Mistry MN, Rossing P, Toto RD, Vart P, Nitsch D, Wheeler DC, Caplin B. Ambient heat exposure and kidney function in patients with chronic kidney disease: a post-hoc analysis of the DAPA-CKD trial. Lancet Planet Health. 2024 Apr;8(4):e225-e233. doi: 10.1016/S2542-5196(24)00026-3. PMID 38580424
- [Derived] Heerspink HJL, Stack AG, Terkeltaub R, Jongs N, Inker LA, Bjursell M, Maklad N, Perl S, Eklund O, Rikte T, Sjostrom CD, Perkovic V; SAPPHIRE Investigators. Combination Treatment with Verinurad and Allopurinol in CKD: A Randomized Placebo and Active Controlled Trial. J Am Soc Nephrol. 2024 May 1;35(5):594-606. doi: 10.1681/ASN.0000000000000326. Epub 2024 Feb 20. PMID 38564654
- [Derived] Koshino A, Schechter M, Chertow GM, Vart P, Jongs N, Toto RD, Rossing P, Correa-Rotter R, McMurray JJV, Gorriz JL, Isidto R, Kashihara N, Langkilde AM, Wheeler DC, Heerspink HJL. Dapagliflozin and Anemia in Patients with Chronic Kidney Disease. NEJM Evid. 2023 Jun;2(6):EVIDoa2300049. doi: 10.1056/EVIDoa2300049. Epub 2023 May 19. PMID 38320128
- [Derived] Yu MK, Vart P, Jongs N, Correa-Rotter R, Rossing P, McMurray JJV, Hou FF, Douthat W, Khullar D, Langkilde AM, Wheeler DC, Heerspink HJL, Chertow GM. Effects of Dapagliflozin in Chronic Kidney Disease Across the Spectrum of Age and by Sex. J Gen Intern Med. 2024 May;39(6):921-930. doi: 10.1007/s11606-023-08397-9. Epub 2023 Dec 14. PMID 38097862
- [Derived] Fletcher RA, Jongs N, Chertow GM, McMurray JJV, Arnott C, Jardine MJ, Mahaffey KW, Perkovic V, Rockenschaub P, Rossing P, Correa-Rotter R, Toto RD, Vaduganathan M, Wheeler DC, Heerspink HJL, Neuen BL. Effect of SGLT2 Inhibitors on Discontinuation of Renin-angiotensin System Blockade: A Joint Analysis of the CREDENCE and DAPA-CKD Trials. J Am Soc Nephrol. 2023 Dec 1;34(12):1965-1975. doi: 10.1681/ASN.0000000000000248. Epub 2023 Oct 25. PMID 37876229
- [Derived] Heerspink HJL, Jongs N, Schloemer P, Little DJ, Brinker M, Tasto C, Karpefors M, Wheeler DC, Bakris G, Perkovic V, Nkulikiyinka R, Rossert J, Gasparyan SB. Development and Validation of a New Hierarchical Composite End Point for Clinical Trials of Kidney Disease Progression. J Am Soc Nephrol. 2023 Dec 1;34(12):2025-2038. doi: 10.1681/ASN.0000000000000243. Epub 2023 Oct 24. PMID 37872654
- [Derived] Chertow GM, Correa-Rotter R, Vart P, Jongs N, McMurray JJV, Rossing P, Langkilde AM, Sjostrom CD, Toto RD, Wheeler DC, Heerspink HJL; DAPA-CKD Trial Committees and Investigators. Effects of Dapagliflozin in Chronic Kidney Disease, With and Without Other Cardiovascular Medications: DAPA-CKD Trial. J Am Heart Assoc. 2023 May 2;12(9):e028739. doi: 10.1161/JAHA.122.028739. Epub 2023 Apr 29. PMID 37119064
- [Derived] Vart P, Jongs N, Wheeler DC, Heerspink HJL, Langkilde AM, Chertow GM. Effectiveness and Safety of Dapagliflozin for Black vs White Patients With Chronic Kidney Disease in North and South America: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e2310877. doi: 10.1001/jamanetworkopen.2023.10877. PMID 37103935
- [Derived] Willigers BJA, Ouwens M, Briggs A, Heerspink HJL, Pollock C, Pecoits-Filho R, Tangri N, Kovesdy CP, Wheeler DC, Garcia Sanchez JJ. The Role of Expert Opinion in Projecting Long-Term Survival Outcomes Beyond the Horizon of a Clinical Trial. Adv Ther. 2023 Jun;40(6):2741-2751. doi: 10.1007/s12325-023-02503-3. Epub 2023 Apr 18. PMID 37071317
- [Derived] Schechter M, Jongs N, Chertow GM, Mosenzon O, McMurray JJV, Correa-Rotter R, Rossing P, Langkilde AM, Sjostrom CD, Toto RD, Wheeler DC, Heerspink HJL. Effects of Dapagliflozin on Hospitalizations in Patients With Chronic Kidney Disease : A Post Hoc Analysis of DAPA-CKD. Ann Intern Med. 2023 Jan;176(1):59-66. doi: 10.7326/M22-2115. Epub 2022 Dec 6. PMID 36469914
- [Derived] Vart P, Vaduganathan M, Jongs N, Remuzzi G, Wheeler DC, Hou FF, McCausland F, Chertow GM, Heerspink HJL. Estimated Lifetime Benefit of Combined RAAS and SGLT2 Inhibitor Therapy in Patients with Albuminuric CKD without Diabetes. Clin J Am Soc Nephrol. 2022 Dec;17(12):1754-1762. doi: 10.2215/CJN.08900722. Epub 2022 Nov 22. PMID 36414316
- [Derived] McEwan P, Darlington O, Miller R, McMurray JJV, Wheeler DC, Heerspink HJL, Briggs A, Bergenheim K, Garcia Sanchez JJ. Cost-Effectiveness of Dapagliflozin as a Treatment for Chronic Kidney Disease: A Health-Economic Analysis of DAPA-CKD. Clin J Am Soc Nephrol. 2022 Dec;17(12):1730-1741. doi: 10.2215/CJN.03790322. Epub 2022 Nov 2. PMID 36323444
- [Derived] Jongs N, Chertow GM, Greene T, McMurray JJV, Langkilde AM, Correa-Rotter R, Kashihara N, Rossing P, Sjostrom CD, Stefansson BV, Toto RD, Wheeler DC, Heerspink HJL; DAPA-CKD Trial Committees and Investigators; Members of the DAPA-CKD Trial Committees and Investigators. Correlates and Consequences of an Acute Change in eGFR in Response to the SGLT2 Inhibitor Dapagliflozin in Patients with CKD. J Am Soc Nephrol. 2022 Nov;33(11):2094-2107. doi: 10.1681/ASN.2022030306. Epub 2022 Aug 17. PMID 35977807
- [Derived] Vart P, Correa-Rotter R, Hou FF, Jongs N, Chertow GM, Langkilde AM, McMurray JJV, Rossing P, Sjostrom CD, Stefansson BV, Toto RD, Douthat W, Escudero E, Isidto R, Khullar D, Bajaj HS, Wheeler DC, Heerspink HJL. Efficacy and Safety of Dapagliflozin in Patients With CKD Across Major Geographic Regions. Kidney Int Rep. 2022 Feb 2;7(4):699-707. doi: 10.1016/j.ekir.2022.01.1060. eCollection 2022 Apr. PMID 35497805
- [Derived] Waijer SW, Vart P, Cherney DZI, Chertow GM, Jongs N, Langkilde AM, Mann JFE, Mosenzon O, McMurray JJV, Rossing P, Correa-Rotter R, Stefansson BV, Toto RD, Wheeler DC, Heerspink HJL. Effect of dapagliflozin on kidney and cardiovascular outcomes by baseline KDIGO risk categories: a post hoc analysis of the DAPA-CKD trial. Diabetologia. 2022 Jul;65(7):1085-1097. doi: 10.1007/s00125-022-05694-6. Epub 2022 Apr 21. PMID 35445820
- [Derived] Heerspink HJL, Jongs N, Chertow GM, Langkilde AM, McMurray JJV, Correa-Rotter R, Rossing P, Sjostrom CD, Stefansson BV, Toto RD, Wheeler DC, Greene T; DAPA-CKD Trial Committees and Investigators. Effect of dapagliflozin on the rate of decline in kidney function in patients with chronic kidney disease with and without type 2 diabetes: a prespecified analysis from the DAPA-CKD trial. Lancet Diabetes Endocrinol. 2021 Nov;9(11):743-754. doi: 10.1016/S2213-8587(21)00242-4. Epub 2021 Oct 4. PMID 34619108
- [Derived] Jongs N, Greene T, Chertow GM, McMurray JJV, Langkilde AM, Correa-Rotter R, Rossing P, Sjostrom CD, Stefansson BV, Toto RD, Wheeler DC, Heerspink HJL; DAPA-CKD Trial Committees and Investigators. Effect of dapagliflozin on urinary albumin excretion in patients with chronic kidney disease with and without type 2 diabetes: a prespecified analysis from the DAPA-CKD trial. Lancet Diabetes Endocrinol. 2021 Nov;9(11):755-766. doi: 10.1016/S2213-8587(21)00243-6. Epub 2021 Oct 4. PMID 34619106
- [Derived] McMurray JJV, Wheeler DC, Stefansson BV, Jongs N, Postmus D, Correa-Rotter R, Chertow GM, Hou FF, Rossing P, Sjostrom CD, Solomon SD, Toto RD, Langkilde AM, Heerspink HJL; DAPA-CKD Trial Committees and Investigators. Effects of Dapagliflozin in Patients With Kidney Disease, With and Without Heart Failure. JACC Heart Fail. 2021 Nov;9(11):807-820. doi: 10.1016/j.jchf.2021.06.017. Epub 2021 Aug 23. PMID 34446370
- [Derived] Persson F, Rossing P, Vart P, Chertow GM, Hou FF, Jongs N, McMurray JJV, Correa-Rotter R, Bajaj HS, Stefansson BV, Toto RD, Langkilde AM, Wheeler DC, Heerspink HJL; DAPA-CKD Trial Committees and Investigators. Efficacy and Safety of Dapagliflozin by Baseline Glycemic Status: A Prespecified Analysis From the DAPA-CKD Trial. Diabetes Care. 2021 Aug;44(8):1894-1897. doi: 10.2337/dc21-0300. Epub 2021 Jun 28. PMID 34183431
- [Derived] Wheeler DC, Stefansson BV, Jongs N, Chertow GM, Greene T, Hou FF, McMurray JJV, Correa-Rotter R, Rossing P, Toto RD, Sjostrom CD, Langkilde AM, Heerspink HJL; DAPA-CKD Trial Committees and Investigators. Effects of dapagliflozin on major adverse kidney and cardiovascular events in patients with diabetic and non-diabetic chronic kidney disease: a prespecified analysis from the DAPA-CKD trial. Lancet Diabetes Endocrinol. 2021 Jan;9(1):22-31. doi: 10.1016/S2213-8587(20)30369-7. PMID 33338413
- [Derived] McMurray JJV, Wheeler DC, Stefansson BV, Jongs N, Postmus D, Correa-Rotter R, Chertow GM, Greene T, Held C, Hou FF, Mann JFE, Rossing P, Sjostrom CD, Toto RD, Langkilde AM, Heerspink HJL; DAPA-CKD Trial Committees and Investigators. Effect of Dapagliflozin on Clinical Outcomes in Patients With Chronic Kidney Disease, With and Without Cardiovascular Disease. Circulation. 2021 Feb 2;143(5):438-448. doi: 10.1161/CIRCULATIONAHA.120.051675. Epub 2020 Nov 13. PMID 33186054
- [Derived] Heerspink HJL, Stefansson BV, Correa-Rotter R, Chertow GM, Greene T, Hou FF, Mann JFE, McMurray JJV, Lindberg M, Rossing P, Sjostrom CD, Toto RD, Langkilde AM, Wheeler DC; DAPA-CKD Trial Committees and Investigators. Dapagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2020 Oct 8;383(15):1436-1446. doi: 10.1056/NEJMoa2024816. Epub 2020 Sep 24. PMID 32970396
- [Derived] Wheeler DC, Stefansson BV, Batiushin M, Bilchenko O, Cherney DZI, Chertow GM, Douthat W, Dwyer JP, Escudero E, Pecoits-Filho R, Furuland H, Gorriz JL, Greene T, Haller H, Hou FF, Kang SW, Isidto R, Khullar D, Mark PB, McMurray JJV, Kashihara N, Nowicki M, Persson F, Correa-Rotter R, Rossing P, Toto RD, Umanath K, Van Bui P, Wittmann I, Lindberg M, Sjostrom CD, Langkilde AM, Heerspink HJL. The dapagliflozin and prevention of adverse outcomes in chronic kidney disease (DAPA-CKD) trial: baseline characteristics. Nephrol Dial Transplant. 2020 Oct 1;35(10):1700-1711. doi: 10.1093/ndt/gfaa234. PMID 32862232
- [Derived] Piperidou A, Loutradis C, Sarafidis P. SGLT-2 inhibitors and nephroprotection: current evidence and future perspectives. J Hum Hypertens. 2021 Jan;35(1):12-25. doi: 10.1038/s41371-020-00393-4. Epub 2020 Aug 10. PMID 32778748
- [Derived] Sternlicht HK, Bakris GL. Reductions in albuminuria with SGLT2 inhibitors: a marker for improved renal outcomes in patients without diabetes? Lancet Diabetes Endocrinol. 2020 Jul;8(7):553-555. doi: 10.1016/S2213-8587(20)30185-6. No abstract available. PMID 32559465
- [Derived] Gonzalez DE, Foresto RD, Ribeiro AB. SGLT-2 inhibitors in diabetes: a focus on renoprotection. Rev Assoc Med Bras (1992). 2020 Jan 13;66Suppl 1(Suppl 1):s17-s24. doi: 10.1590/1806-9282.66.S1.17. PMID 31939531
- See also: redacted protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D169AC00001&attachmentIdentifier=c59c2c03-ebfa-46f4-beac-d0b14b62db99&fileName=d169ac00001_csp_Redacted.pdf&versionIdentifier=
- See also: redacted Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D169AC00001&attachmentIdentifier=987ded9e-acd7-4718-a380-431a2b2d1377&fileName=d169ac00001_sap_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapagliflozin: Dapagliflozin 10 mg, given once daily per oral use
- Placebo: Placebo tablet to match dapagliflozin 10 mg, given once daily per oral use
Period: Overall Study
Arm/Group | Dapagliflozin | Placebo
Started | 2152 | 2152
Completed | 2142 | 2147
Not Completed | 10 | 5
Not completed — Withdrawal by Subject | 8 | 3
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 2152 | 2152 | 4304
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (12.1) | 61.9 (12.1) | 61.8 (12.1)
Age, Customized [Count of Participants; unit: Participants]
  <= 50 years | 362 | 370 | 732
  > 50 years | 1790 | 1782 | 3572
Age, Customized [Count of Participants; unit: Participants]
  <= 65 years | 1247 | 1239 | 2486
  > 65 years | 905 | 913 | 1818
Age, Customized [Count of Participants; unit: Participants]
  <=65 years | 1247 | 1239 | 2486
  66-75 years | 663 | 667 | 1330
  > 75 years | 242 | 246 | 488
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 709 | 716 | 1425
  Male | 1443 | 1436 | 2879
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 522 | 550 | 1072
  Not Hispanic or Latino | 1630 | 1602 | 3232
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1124 | 1166 | 2290
  Black or African American | 104 | 87 | 191
  Asian | 749 | 718 | 1467
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  American Indian or Alaska Native | 62 | 74 | 136
  Other | 112 | 106 | 218
Most likely etiology of CKD [Count of Participants; unit: Participants]
  Diabetic Nephropathy | 1271 | 1239 | 2510
  Ischaemic/Hypertensive Nephropathy | 324 | 363 | 687
  Chronic Glomerulonephritis | 343 | 352 | 695
  Other or unknown cause of CKD | 214 | 198 | 412
eGFR [Mean (Standard Deviation); unit: mL/min/1.73 m2] | 43.2 (12.3) | 43.0 (12.4) | 43.1 (12.4)
Urine albumin creatinine ratio [Median (Inter-Quartile Range); unit: mg/g] | 965 [472 to 1903] | 934 [482 to 1869] | 949 [477 to 1865]
Type 2 Diabetes Mellitus at Baseline [Count of Participants; unit: Participants]
  Yes | 1455 | 1451 | 2906
  No | 697 | 701 | 1398

OUTCOME MEASURES:

1. Primary Outcome: Time to the First Occurrence of Any of the Components of the Composite: ≥50% Sustained Decline in eGFR or Reaching ESRD or CV Death or Renal Death.
Description: End Stage Renal Disease (ESRD) is defined as:
  * Sustained eGFR <15 mL/min/1.73m2 or,
  * Chronic dialysis treatment or,
  * Receiving a renal transplant The proportional hazards Cox regression model takes into account the time to the event. Data is reported as the numbers of subjects with the event and the Hazard ratio is included in the Statistical Analysis section attached to the Outcome Measure data table.
Time Frame: Up to 38.2 months
Population: For the primary endpoint the Full Analysis Set was used. This included all patients who were randomized to study treatment. Patients were analyzed according to their randomized treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 2152 | 2152
Participants | 197 | 312
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority; p < 0.0001, Regression, Cox; Stratified by randomization stratification of Type 2 Diabetes and urine albumin creatinine ratio and adjusting for baseline eGFR; Hazard Ratio (HR) = 0.61, 95% CI [0.51 to 0.72]

2. Secondary Outcome: Time to the First Occurrence of Any of the Components of the Composite: ≥50% Sustained Decline in eGFR or Reaching ESRD or Renal Death.
Description: as for outcome 1
Time Frame: Up to 38.2 months
Population: For the secondary endpoints the Full Analysis Set was used. This included all patients who were randomized to study treatment. Patients were analyzed according to their randomized treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 2152 | 2152
Participants | 142 | 243
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority; p < 0.0001, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.56, 95% CI [0.45 to 0.68]

3. Secondary Outcome: Time to the First Occurrence of Either of the Components of the Composite: CV Death or Hospitalization for Heart Failure.
Description: The proportional hazards Cox regression model takes into account the time to the event. Data is reported as the numbers of subjects with the event and the Hazard ratio is included in the Statistical Analysis section attached to the Outcome Measure data table.
Time Frame: Up to 38.2 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 2152 | 2152
Participants | 100 | 138
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority; p = 0.0089, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.71, 95% CI [0.55 to 0.92]

4. Secondary Outcome: Time to Death From Any Cause.
Description: as for outcome 3
Time Frame: Up to 38.2 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 2152 | 2152
Participants | 101 | 146
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Superiority; p = 0.0035, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.69, 95% CI [0.53 to 0.88]

ADVERSE EVENTS:
Time Frame: Up to 39.2 months
Description: For All Cause Mortality, the Full Analysis Set was used. This included all patients who were randomized to study drug. For analysis of Serious Adverse Events, Safety analysis set was used. Safety analysis set consisted of all randomized patients who received at least one dose of study drug.
Groups:
- Dapa 10 mg: Dapagliflozin 10 mg, given once daily per oral use
Arm/Group | Dapa 10 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 107/2152 | 159/2152
Serious Adverse Events (participants affected / at risk) | 633/2149 | 729/2149
Other Adverse Events (participants affected / at risk) | 479/2149 | 500/2149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapa 10 mg (N=2149) | Placebo (N=2149)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 8 (8)
Blood loss anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (3)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 6 (6)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 2 (2)
Acute left ventricular failure (Cardiac disorders) | 5 (5) | 10 (12)
Acute myocardial infarction (Cardiac disorders) | 32 (35) | 46 (56)
Angina pectoris (Cardiac disorders) | 4 (5) | 9 (9)
Angina unstable (Cardiac disorders) | 14 (17) | 22 (26)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 8 (8) | 17 (18)
Atrial flutter (Cardiac disorders) | 1 (1) | 3 (3)
Atrioventricular block (Cardiac disorders) | 2 (2) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 3 (3) | 5 (5)
Atrioventricular block second degree (Cardiac disorders) | 2 (2) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 3 (3) | 3 (3)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 4 (4) | 10 (10)
Cardiac failure (Cardiac disorders) | 39 (56) | 59 (72)
Cardiac failure acute (Cardiac disorders) | 4 (5) | 7 (8)
Cardiac failure chronic (Cardiac disorders) | 3 (4) | 5 (5)
Cardiac failure congestive (Cardiac disorders) | 13 (17) | 22 (29)
Cardio-respiratory arrest (Cardiac disorders) | 5 (5) | 3 (4)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 2 (2)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 4 (4) | 10 (10)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 3 (3)
Defect conduction intraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 3 (5)
Ischaemic cardiomyopathy (Cardiac disorders) | 4 (4) | 4 (4)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 11 (11) | 6 (7)
Myocardial ischaemia (Cardiac disorders) | 6 (6) | 6 (7)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Vestibular disorder (Ear and labyrinth disorders) | 5 (7) | 3 (3)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Hyperadrenocorticism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0)
Pituitary-dependent cushing's syndrome (Endocrine disorders) | 0 (0) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 8 (12) | 6 (8)
Cataract subcapsular (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 4 (4) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Ocular ischaemic syndrome (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 3 (3)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vitreous disorder (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Diverticular perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 3 (4)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 2 (2)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3) | 5 (6)
Gastritis hypertrophic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 6 (7)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric vascular insufficiency (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Palatal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 5 (6) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 1 (1)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 4 (4)
Varices oesophageal (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 2 (3)
Cardiac death (General disorders) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 3 (3)
Death (General disorders) | 15 (15) | 27 (27)
Fatigue (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 3 (3)
Impaired healing (General disorders) | 1 (1) | 2 (2)
Inflammation (General disorders) | 2 (2) | 0 (0)
Medical device site discomfort (General disorders) | 0 (0) | 1 (1)
Medical device site pain (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 5 (5)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 4 (4)
Stent-graft endoleak (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 2 (2)
Sudden death (General disorders) | 4 (4) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 4 (4) | 4 (4)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 5 (5)
Cholecystitis chronic (Hepatobiliary disorders) | 2 (2) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (2) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1)
Acquired immunodeficiency syndrome (Infections and infestations) | 1 (1) | 0 (0)
Acute hepatitis b (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 3 (3)
Appendicitis (Infections and infestations) | 3 (3) | 3 (3)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 2 (2)
Bacteraemia (Infections and infestations) | 3 (3) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 2 (2)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 5 (5) | 6 (7)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 14 (17) | 15 (20)
Cellulitis gangrenous (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 4 (5) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Dengue haemorrhagic fever (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 1 (1)
Device related sepsis (Infections and infestations) | 2 (2) | 0 (0)
Diabetic foot infection (Infections and infestations) | 5 (8) | 5 (6)
Diabetic gangrene (Infections and infestations) | 2 (2) | 2 (2)
Diverticulitis (Infections and infestations) | 5 (5) | 5 (5)
Empyema (Infections and infestations) | 1 (1) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 3 (3) | 5 (6)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Fournier's gangrene (Infections and infestations) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Fungal oesophagitis (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 1 (1)
Gangrene (Infections and infestations) | 7 (7) | 3 (4)
Gas gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 10 (11) | 9 (9)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 4 (4)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
Infected skin ulcer (Infections and infestations) | 2 (3) | 2 (3)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 3 (3)
Inguinal hernia gangrenous (Infections and infestations) | 0 (0) | 1 (1)
Intestinal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Leishmaniasis (Infections and infestations) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 3 (4) | 0 (0)
Localised infection (Infections and infestations) | 3 (3) | 8 (8)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Mastoiditis (Infections and infestations) | 1 (1) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Meningoencephalitis herpetic (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 10 (12) | 12 (13)
Osteomyelitis chronic (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 2 (2) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 2 (2)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1)
Plasmodium falciparum infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 44 (50) | 70 (79)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (2) | 3 (3)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 5 (5) | 2 (2)
Pyonephrosis (Infections and infestations) | 1 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Rocky mountain spotted fever (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 13 (13) | 18 (18)
Septic shock (Infections and infestations) | 11 (11) | 11 (11)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 1 (1)
Splenic abscess (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Superinfection viral (Infections and infestations) | 0 (0) | 1 (1)
Suspected covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Tuberculosis bladder (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 20 (22) | 15 (21)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urogenital infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 4 (4) | 3 (3)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulval cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 7 (7) | 4 (5)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Inflammation of wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lenticular injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 5 (5) | 1 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Vascular access malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood parathyroid hormone increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Fibrin d dimer increased (Investigations) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 2 (2) | 3 (3)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 7 (9)
Diabetes mellitus (Metabolism and nutrition disorders) | 9 (11) | 5 (6)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Gout (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (8) | 17 (19)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (6) | 12 (12)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 9 (9) | 18 (19)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Milk-alkali syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Shock hypoglycaemic (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Benign biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Bone giant cell tumour malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Epithelioid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 2 (2)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 6 (6)
Lymphoplasmacytoid lymphoma/immunocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Peripheral t-cell lymphoma unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 6 (6)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Prostate cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cell carcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal hamartoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Testicular germ cell cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Brain hypoxia (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 6 (6) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 8 (8) | 3 (4)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral vasoconstriction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 10 (10) | 8 (8)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 2 (2) | 0 (0)
Diabetic hyperosmolar coma (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (1) | 4 (4)
Facial nerve disorder (Nervous system disorders) | 2 (2) | 0 (0)
Facial paralysis (Nervous system disorders) | 2 (2) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 3 (3) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 22 (23) | 28 (29)
Lacunar stroke (Nervous system disorders) | 2 (2) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Motor neurone disease (Nervous system disorders) | 1 (1) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Putamen haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 7 (7) | 5 (5)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 11 (11) | 9 (10)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 2 (2)
Device power source issue (Product Issues) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 4 (4)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Post stroke depression (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 39 (43) | 52 (64)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 20 (24) | 31 (34)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 2 (2) | 3 (3)
End stage renal disease (Renal and urinary disorders) | 26 (27) | 36 (39)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerulonephritis chronic (Renal and urinary disorders) | 2 (3) | 6 (9)
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 0 (0) | 2 (6)
Haematuria (Renal and urinary disorders) | 3 (4) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (2) | 1 (1)
Iga nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Intercapillary glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 4 (4)
Nephropathy (Renal and urinary disorders) | 2 (2) | 3 (3)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 4 (4)
Nephrosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 3 (5)
Obstructive nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 3 (4)
Renal amyloidosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 6 (6) | 10 (11)
Renal impairment (Renal and urinary disorders) | 14 (15) | 15 (15)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urate nephropathy (Renal and urinary disorders) | 0 (0) | 1 (3)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urethral dilatation (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 4 (4)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Vesical fistula (Renal and urinary disorders) | 0 (0) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 6 (6) | 4 (4)
Endometrial disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Seminal vesicular cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 11 (12)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 10 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (8)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (10)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (7)
Aortic aneurysm (Vascular disorders) | 0 (0) | 2 (2)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 2 (2)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 6 (6) | 6 (6)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 3 (3) | 0 (0)
Femoral artery embolism (Vascular disorders) | 1 (1) | 0 (0)
Granulomatosis with polyangiitis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 9 (13) | 10 (10)
Hypertensive crisis (Vascular disorders) | 6 (6) | 5 (5)
Hypertensive emergency (Vascular disorders) | 0 (0) | 6 (7)
Hypertensive urgency (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 8 (8) | 3 (3)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery embolism (Vascular disorders) | 1 (1) | 0 (0)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 6 (8) | 7 (7)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 3 (3) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (2) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 4 (4) | 8 (8)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapa 10 mg (N=2149) | Placebo (N=2149)
Diarrhoea (Gastrointestinal disorders) | 45 (56) | 41 (46)
Oedema peripheral (General disorders) | 54 (56) | 63 (75)
Nasopharyngitis (Infections and infestations) | 92 (136) | 81 (118)
Urinary tract infection (Infections and infestations) | 78 (102) | 79 (96)
Glomerular filtration rate decreased (Investigations) | 39 (45) | 61 (67)
Hyperkalaemia (Metabolism and nutrition disorders) | 53 (67) | 49 (54)
Hypoglycaemia (Metabolism and nutrition disorders) | 74 (119) | 70 (96)
Back pain (Musculoskeletal and connective tissue disorders) | 44 (46) | 50 (52)
Acute kidney injury (Renal and urinary disorders) | 49 (54) | 44 (50)
Renal impairment (Renal and urinary disorders) | 51 (55) | 64 (72)
Hypertension (Vascular disorders) | 62 (63) | 60 (66)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT03036150/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT03036150/SAP_001.pdf